CLINICAL TRIAL: NCT00639860
Title: Clinical and Histological Evaluation of OSSIX-Plus Resorbable Collagen Membranes for Alveolar Ridge Preservation Following Exodontia
Brief Title: Evaluation of OSSIX-Plus Resorbable Collagen Membranes for Alveolar Ridge Preservation Following Exodontia
Acronym: OSSIX
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: William Giannobile (Other)
Collaborators: Johnson & Johnson (Industry); OraPharma (Industry)
Responsible Party: Sponsor-Investigator, William Giannobile, William Giannobile, D.D.S., D.Med.Sc., University of Michigan
Organization: University of Michigan (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HUM00016574
Record Dates: First submitted 2008-03-14; First posted 2008-03-20 (Estimated); Results first posted 2016-03-31 (Estimated); Last update posted 2016-03-31 (Estimated); Status verified 2016-03

CONDITIONS: Alveolar Bone Loss; Loss of Teeth Due to Extraction; Edentulous Alveolar Ridge
Keywords: extraction; implant; alveolar ridge preservation
MeSH Terms: conditions — Alveolar Bone Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Placing OSSIX-Plus in Extraction Site (Experimental): Placement of OSSIX-Plus, a resorbable collagen membrane, and the promotion of bone healing following exodontia.
  Interventions: Device: OSSIX-Plus

INTERVENTIONS:
Device: OSSIX-Plus — resorbable collagen membrane

SUMMARY:
The purpose of this study is to evaluate clinically, histologically and radiographically the healing of extraction sockets covered with a resorbable collagen membrane (OSSIX-Plus) 12 weeks following exodontia.

DETAILED DESCRIPTION:
Reduction in alveolar ridge height and width may prohibit optimal implant placement, and often compromises the esthetic and functional result. Alveolar ridge preservation has been evaluated in many studies. A variety of bone grafting materials and barrier membranes have been studied for their ability to enhance bone formation in damaged alveolar ridges, and to evaluate their bone healing and bone-forming capacity in extraction sockets. However, the newly developed resorbable collagen membrane OSSIX-Plus has not been evaluated for this purpose. This study is designed to test the ability of OSSIX-Plus (OraPharma Inc., Warminster, Pennsylvania) in promoting optimal bone healing following exodontia. We hypothesize that use of OSSIX-Plus will result in preservation of the height, width and density of the residual alveolar ridge following tooth extraction.

ELIGIBILITY:
Inclusion Criteria:

* Systemically healthy subjects with 1 maxillary premolar tooth requiring extraction
* Residual extraction sockets must have < 80% bone loss in all dimensions (3 or 4-walled bony defects)
* Nonsmokers (individuals who quit smoking at least 6 months prior to the study will be allowed to participate)
* Subjects willing and able to comply with all study-related procedures including maintenance of good oral hygiene and compliance with re-evaluation appointments
* Subjects who read, understand and are willing to sign an informed consent statement

Exclusion Criteria:

* Inadequate zone of keratinized gingiva (KG) or alveolar mucosa to obtain primary wound closure of the surgical site
* Presence of acute infections at the time of tooth extraction
* Clinically significant or unstable (as defined by the investigators) systemic diseases affecting bone or soft tissue growth or other renal, hepatic, cardiac, endocrine, hematological, autoimmune or acute infectious diseases that makes interpretation of the data more difficult
* History of head & neck radiation therapy
* Subjects taking steroids, tetracycline or tetracycline analogs, bone therapeutic levels of fluorides, biphosphonatesm, medications affecting bone turnover, antibiotics for > 7 days or any investigational drug
* Patients who are or become pregnant during the length of the study
* Sites in which one or both adjacent teeth are missing

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2008-03; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William V Giannobile, DDS, DMedSc, Principal Investigator — Professor
Locations (1):
- Michigan Center for Oral Health Research, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Neiva R, Pagni G, Duarte F, Park CH, Yi E, Holman LA, Giannobile WV. Analysis of tissue neogenesis in extraction sockets treated with guided bone regeneration: clinical, histologic, and micro-CT results. Int J Periodontics Restorative Dent. 2011 Sep-Oct;31(5):457-69. PMID 21845241

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placing OSSIX-Plus in Extraction Site
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Placing OSSIX-Plus in Extraction Site
Number analyzed (Participants) | 10
Age, Customized [Median (Full Range); unit: years] | 47.7 [25 to 64]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 4
Region of Enrollment [Number; unit: participants]
  United States | 10
Socket width (buccopalatal) [Mean (Full Range); unit: mm] | 8.3 [7.0 to 10.0]
Socket width (meiodistal) [Mean (Full Range); unit: mm] | 5.1 [4.0 to 8.0]
Stent to buccal plate [Mean (Full Range); unit: mm] | 5.6 [4.0 to 8.0]
Stent to mesial osseous crest [Mean (Full Range); unit: mm] | 4.0 [2.0 to 6.0]
Stent to distal osseous crest [Mean (Full Range); unit: mm] | 4.1 [2.0 to 6.0]
Stent to midosseous crest [Mean (Full Range); unit: mm] | 4.7 [3.0 to 7.0]
Stent to apex of socket [Median (Full Range); unit: mm] | 16.5 [11.0 to 20.0]

OUTCOME MEASURES:

1. Primary Outcome: Change in Bone Gain or Loss in Millimeters (Buccopalatal)
Description: Socket width (buccopalatal) measured by a calibrated examiner using a University of North Carolina (UNC) probe.
Time Frame: From Baseline to 12 weeks
Measure: Mean (Full Range); unit: mm
Arm/Group | Placing OSSIX-Plus in Extraction Site
Number analyzed (Participants) | 10
mm | 7.7 [0.0 to 10.0]

2. Primary Outcome: Change in Bone Gain or Loss in Millimeters (Mesiodistal)
Description: Socket width (mesiodistal) measured by a calibrated examiner using a University of North Carolina (UNC) probe.
Time Frame: From Baseline to 12 weeks
Measure: Mean (Full Range); unit: mm
Arm/Group | Placing OSSIX-Plus in Extraction Site
Number analyzed (Participants) | 10
mm | 4.6 [0.0 to 8.0]

3. Primary Outcome: Change in Bone Gain or Loss in Millimeters (Stent to Apex)
Description: Stent to apex of socket measured by a calibrated examiner using a University of North Carolina (UNC) probe.
Time Frame: From Baseline to 12 weeks
Measure: Mean (Full Range); unit: mm
Arm/Group | Placing OSSIX-Plus in Extraction Site
Number analyzed (Participants) | 10
mm | 10.9 [3.0 to 20.0]

4. Primary Outcome: Radiographic Bone Changes
Description: Radiographic measures were accomplished utilizing a real-time subtraction program, Computer Assisted Radiographic Evaluation (C.A.R.E.).
Time Frame: From Baseline to 12 weeks
Measure: Mean (Full Range); unit: percentage of bone fill
Arm/Group | Placing OSSIX-Plus in Extraction Site
Number analyzed (Participants) | 10
percentage of bone fill | 86.5 [0 to 100]

5. Primary Outcome: New Bone Formation
Description: Percentage of new bone formation of the alveolar bone core biopsies.
Time Frame: From Baseline to 12 weeks
Measure: Mean (Full Range); unit: percentage of vital bone
Arm/Group | Placing OSSIX-Plus in Extraction Site
Number analyzed (Participants) | 10
percentage of vital bone | 46.09 [0 to 100]

ADVERSE EVENTS:
Arm/Group | Placing OSSIX-Plus in Extraction Site
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No